CLINICAL TRIAL: NCT05045742
Title: Prediction of Patient Deterioration Using Machine Learning
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Biofourmis Inc. (Industry)
Responsible Party: Principal Investigator, David Levine, Attending Physician, Brigham and Women's Hospital
Other Study IDs: 2017P002583d
Record Dates: First submitted 2021-04-14; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Infection; Heart Failure; Chronic Obstructive Pulmonary Disease; Asthma; Gout Flare; Chronic Kidney Diseases; Hypertensive Urgency; Atrial Fibrillation Rapid; Anticoagulants; Increased
MeSH Terms: conditions — Infections; Heart Failure; Pulmonary Disease, Chronic Obstructive; Asthma; Renal Insufficiency, Chronic; Hypertensive Crisis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training: A subset of patients that are used to train the machine learning algorithm.
  Interventions: Other: Traditional vital sign alarms versus the BioVitals Index vs the National Early Warning Score 2
- Validation: A subset of patients that are "held back" and used to validate the algorithm's accuracy.
  Interventions: Other: Traditional vital sign alarms versus the BioVitals Index vs the National Early Warning Score 2

INTERVENTIONS:
Other: Traditional vital sign alarms versus the BioVitals Index vs the National Early Warning Score 2 — We will retrospectively compare the alarms produced from traditional vital sign alarms (thresholds set by clinicians) versus the BioVitals Index vs the National Early Warning Score 2

SUMMARY:
This is a retrospective observational study drawing on data from the Brigham and Women's Home Hospital database. Sociodemographic and clinic data from a training cohort were used to train a machine learning algorithm to predict patient deterioration throughout a patient's admission. This algorithm was then validated in a validation cohort.

ELIGIBILITY:
Inclusion Criteria:

Cared for in the Brigham and Women's Home Hospital study

Exclusion Criteria:

Incomplete continuous monitoring data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects admitted at Brigham and Women's Hospital and Brigham and Women's Faulkner Hospital who meet primary diagnosis, age, and geographic residence requirements and are enrolled in home hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Alarm burden | From admission to discharge, measured in hours, on average 5 days
  The number of alarms fired per patient per hour

SECONDARY OUTCOMES:
Sensitivity for recognition of a safety composite | From admission to discharge, on average 5 days
  The sensitivity (true positives divided by condition positives) for detection of a safety composite (overnight visit, extra unplanned visit, transfer back to the hospital, death during admission, delirium, loss of consciousness, or other major event).
Specificity for recognition of a safety composite | From admission to discharge, on average 5 days
  The specificity (true negatives divided by condition negatives) for detection of a safety composite (overnight visit, extra unplanned visit, transfer back to the hospital, death during admission, delirium, loss of consciousness, or other major event).
Positive predictive value for recognition of a safety composite | From admission to discharge, on average 5 days
  The positive predictive value (true positives divided by the sum of true positives plus false positives) for detection of a safety composite (overnight visit, extra unplanned visit, transfer back to the hospital, death during admission, delirium, loss of consciousness, or other major event).
Negative predictive value for recognition of a safety composite | From admission to discharge, on average 5 days
  The negative predictive value (true negatives divided by the sum of true negatives plus false negatives) for detection of a safety composite (overnight visit, extra unplanned visit, transfer back to the hospital, death during admission, delirium, loss of consciousness, or other major event).
Rate of alarms with clinical utility | From admission to discharge, on average 5 days
  We will use general estimating equations (GEE) with three outcomes per patient (the number of clinically important alarms for BioVitals, NEWS2, and traditional vital signs); the GEE will account for the clustering between the three outcomes on a patient. The GEE will use a negative binomial marginal model with a log-link for the number of alarms with clinical utility and an offset for log length-of stay (in hours); with this model, we model the rate per hour of number of alarms with clinical utility with BI, NEWS2, and traditional vital signs. The main covariate in the negative binomial model will be a three-level covariate for method: BI vs NEWS2 vs traditional vital signs, and the exponential of the effect of this covariate will be a pair-wise rate ratio for BI vs NEWS2 vs traditional vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: David Levine, MD MPH MA, Principal Investigator — Associate Physician
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Faulkner Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No